CLINICAL TRIAL: NCT00762554
Title: A Comparison of Single Dose Depodur With Fentanyl Infusion for Post-Cesarean Section Analgesia
Brief Title: Depodur vs Fentanyl Infusion for Post-C/S Analgesia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Uncertain safety of one of the study medications.
Sponsor: Goodman, Evan, M.D. (Individual)
Responsible Party: Principal Investigator, Dr. Evan Goodman, MD, Anesthesiologist, Goodman, Evan, M.D.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: goodman-1
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Analgesia
Keywords: analgesia; cesarean section; fentanyl; Depodur; Post-cesarean section analgesia
MeSH Terms: conditions — Agnosia | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Epidural Depodur after spinal bupivacaine
  Interventions: Drug: Depodur
- 2 (Active Comparator): Epidural fentanyl infusion after epidural lidocaine or spinal bupivacaine
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Depodur — Depodur 10mg given epidurally at end of cesarean section.
  Arms: 1
Drug: Depodur — Depodur 10mg given epidurally at end of cesarean section after patient received spinal bupivacaine at the beginning of the case.
  Arms: 1
Drug: Fentanyl — Epidural fentanyl infusion started after spinal bupivacaine used for the cesarean section.
  Arms: 2

SUMMARY:
Epidurally administered Depodur provides equal or superior analgesia as an epidural infusion of fentanyl for the first 48 hours after a cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women (ASA I or II) who are scheduled for an elective cesarean section
* Patient appropriate for regional anesthesia
* Patient agrees to receive regional anesthesia
* Patient willing to have an epidural infusion of medication for two days postoperatively

Exclusion Criteria:

* Morbid obesity
* History of sleep apnea
* Allergy to opioids medications
* History of opioids use during week prior to procedure
* Emergency cesarean section
* Significant surgical complications
* Contraindication or refusal to have regional anesthesia
* Age less than 18

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Degree of analgesia (measured on a 10-point scale) | 48 hours post-operatively

SECONDARY OUTCOMES:
Frequency of minor side effects, such as pruritis or nausea. | 48 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Carvalho B, Riley E, Cohen SE, Gambling D, Palmer C, Huffnagle HJ, Polley L, Muir H, Segal S, Lihou C, Manvelian G; DepoDur Study Group. Single-dose, sustained-release epidural morphine in the management of postoperative pain after elective cesarean delivery: results of a multicenter randomized controlled study. Anesth Analg. 2005 Apr;100(4):1150-1158. doi: 10.1213/01.ANE.0000149544.58230.FF. PMID 15781537
- [Background] Carvalho B, Roland LM, Chu LF, Campitelli VA 3rd, Riley ET. Single-dose, extended-release epidural morphine (DepoDur) compared to conventional epidural morphine for post-cesarean pain. Anesth Analg. 2007 Jul;105(1):176-83. doi: 10.1213/01.ane.0000265533.13477.26. PMID 17578973